CLINICAL TRIAL: NCT00285844
Title: Integrating the Genetic and Metabolic Faces of Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RDK071309
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Insulin Resistance; Obesity; Metabolic Syndrome
Keywords: obesity; insulin resistance; thiazolidinedione; weight loss; adipose tissue; metabolic syndrome; diabetes prevention; cardiovascular disease prevention
MeSH Terms: conditions — Insulin Resistance; Obesity; Metabolic Syndrome; Weight Loss | interventions — 2,4-thiazolidinedione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pioglitazone (Experimental): IR and IS subjects will be randomized to pioglitazone 45 mg daily for 16 wks for comparison with dietary weight loss intervention
  Interventions: Drug: thiazolidinedione
- Dietary Weight Loss (Experimental): IR and IS subjects will be randomized to dietary weight loss for 16 wks for comparison to pioglitazone intervention
  Interventions: Behavioral: weight loss

INTERVENTIONS:
Behavioral: weight loss
  Arms: Dietary Weight Loss
Drug: thiazolidinedione
  Arms: pioglitazone

SUMMARY:
The goal of this study is to determine why some obese individuals develop insulin resistance and others do not. We hypothesize that an impairment in differentiation of fat cells (adipocytes) is responsible for the development of insulin resistance in select obese individuals. This study will evaluate obese individuals at baseline with respect to characteristics of adipocytes, including gene expression, and will then entail randomizing subjects to either weight loss or treatment with an insulin sensitizing drug (pioglitazone). Changes in insulin resistance will be associated with changes in adipocyte morphology and gene expression.

DETAILED DESCRIPTION:
Healthy overweight/obese individuals will be screened for insulin resistance. Both insulin resistant individuals and insulin sensitive individuals (to serve as controls) will be eligible to enroll. Fat cel biopsy and CT scan of the abdomen is required at baseline and after an intervention with either weight loss or pioglitazone (drug to improve insulin resistance). Subjects will repeat insulin resistance test after the intervention as well. Subjects will learn much about their metabolism in this study, and will have an opportunity to improve their insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* nondiabetic defined as fasting plasma glucose < 126 mg/dL
* body mass index 27 to 35 kg/m2
* no major organ diseases
* able to come to Stanford for regular clinical research center visits
* English speaking or has own translator

Exclusion Criteria:

* pregnancy/lactation
* history of eating disorder or major psychiatric illness
* allergy to thiazolidinedione
* elevation of liver enzymes (> 2.5 times upper normal limit)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Adipose Cell Size Distribution | 2005-2012

SECONDARY OUTCOMES:
Adipose Tissue Gene Expression | 2005-2013

OTHER OUTCOMES:
Insulin-Mediated Glucose Uptake | 2005-2012

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, MS, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLaughlin T, Liu LF, Lamendola C, Shen L, Morton J, Rivas H, Winer D, Tolentino L, Choi O, Zhang H, Hui Yen Chng M, Engleman E. T-cell profile in adipose tissue is associated with insulin resistance and systemic inflammation in humans. Arterioscler Thromb Vasc Biol. 2014 Dec;34(12):2637-43. doi: 10.1161/ATVBAHA.114.304636. Epub 2014 Oct 23. PMID 25341798
- [Derived] McLaughlin T, Lamendola C, Liu A, Abbasi F. Preferential fat deposition in subcutaneous versus visceral depots is associated with insulin sensitivity. J Clin Endocrinol Metab. 2011 Nov;96(11):E1756-60. doi: 10.1210/jc.2011-0615. Epub 2011 Aug 24. PMID 21865361
- [Derived] McLaughlin T, Deng A, Yee G, Lamendola C, Reaven G, Tsao PS, Cushman SW, Sherman A. Inflammation in subcutaneous adipose tissue: relationship to adipose cell size. Diabetologia. 2010 Feb;53(2):369-77. doi: 10.1007/s00125-009-1496-3. Epub 2009 Oct 9. PMID 19816674
- [Derived] McLaughlin T, Deng A, Gonzales O, Aillaud M, Yee G, Lamendola C, Abbasi F, Connolly AJ, Sherman A, Cushman SW, Reaven G, Tsao PS. Insulin resistance is associated with a modest increase in inflammation in subcutaneous adipose tissue of moderately obese women. Diabetologia. 2008 Dec;51(12):2303-8. doi: 10.1007/s00125-008-1148-z. Epub 2008 Sep 30. PMID 18825363